CLINICAL TRIAL: NCT03104218
Title: Transcranial Direct Current Stimulation to Enhance Rehabilitation in Individuals With Rotator Cuff Tendinopathy: a Triple-blind Randomized Control Trial
Brief Title: Transcranial Direct Current Stimulation to Enhance Rehabilitation in Individuals With Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Jean-Sébastien Roy
Record Dates: First submitted 2017-02-08; First posted 2017-04-07 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Rotator Cuff Tendinopathy

STUDY DESIGN:
Intervention Model Description: This triple-blind (patients, therapist & evaluator), parallel-group RCT will include four evaluation sessions over 3 months (baseline, week 3, week 6, 3-month) and 8 supervised physiotherapy treatments during a 6-week rehabilitation program (3 sessions the 1st week, 2 sessions the 2nd weeks, 3 session in the last 4 weeks). Thereafter, participants will be randomly assigned to one of two intervention groups, and then take part in their assigned 6-week intervention. At week 3, 6, and 12, the self-administered questionnaires will be re-administered, while US measurements will only be re-evaluated at week 6.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A randomisation list will be established prior to the initiation of the study using a random number generator. The randomisation list will be generated by an independent research assistant not involved in data collection. Allocation will be concealed in sealed and opaque envelopes that will be sequentially numbered. Randomisation will be stratified to ensure balance of the treatment groups with respect to sex. A blocked randomisation will also be used to make sure that two equal groups of 20 participants are obtained. Given that it is possible to blind the treating PT, the participants and the evaluators, a triple-blind design will be used. An independent research assistant from the CIRRIS will open the randomisation envelope indicating the participant's assignment. The research assistant will be blind to the baseline evaluation results. The research assistant will be the one who will set-up the parameters on the tDCS before treatment sessions with tDCS (real or sham tDCS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Experimental): tDCS will be delivered using a direct current stimulator (constant current of 1.5 mA) via two 35cm2 (5 x 7 cm) saline-soaked surface sponge electrodes (parameters shown effective to enhance training). The center of the active electrode will be positioned over C3/C4 (international 10-20 EEG system; corresponding to the cortical representation of upper limb muscles), contralateral to the side of pain and the reference electrode over the contralateral supraorbital region. Current intensity will be ramped up (0-1.5 mA) and down (1.5-0 mA) over 15 seconds at the beginning and end of the 30 minutes stimulation period.
  Interventions: Other: tDCS group
- Placebo group (Sham Comparator): The sham tDCS involves electrodes placed in an identical position to that used for active stimulation; however the stimulation will be turned on for 15 seconds and then off to provide participants with the initial "itching" sensation but without current for the remainder of the period. This procedure has been shown to effectively blind participants to the stimulation condition. The parameters on the tDCS will be set-up by a research assistant before each session. The treating physiotherapist will not have access to the control board of the tDCS.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: tDCS group — Interventions: movement training, strengthening, patient education. tDCS will be delivered using a direct current stimulator (constant current of 1.5 mA) via two 35cm2 (5 x 7 cm) saline-soaked surface sponge electrodes (parameters shown effective to enhance training).40 The center of the active electrode will be positioned over C3/C4 (international 10-20 EEG system; corresponding to the cortical representation of upper limb muscles)57, contralateral to the side of pain and the reference electrode over the contralateral supraorbital region. Current intensity will be ramped up (0-1.5 mA) and down (1.5-0 mA) over 15 seconds at the beginning and end of the 30 minutes stimulation period.
  Arms: tDCS group
Other: Placebo group — Interventions: movement training, strengthening, patient education. The sham tDCS involves electrodes placed in an identical position to that used for active stimulation; however the stimulation will be turned on for 15 seconds and then off to provide participants with the initial "itching" sensation but without current for the remainder of the period. This procedure has been shown to effectively blind participants to the stimulation condition.
  Arms: Placebo group

SUMMARY:
Transcranial direct current stimulation (tDCS), an electrostimulation technique known to modulate the motor cortex excitability, has been shown to enhance the effects of rehabilitation in populations with neurological injuries. tDCS could similarly be effective in individuals with rotator cuff (RC) tendinopathy, as this pathology is also associated with pain and motor control deficits. For the treatment of RC tendinopathy, sensorimotor training is effective to reduce pain, increase function and enhance motor control of the shoulder. The addition of tDCS during sensorimotor training could enhance motor learning associated with sensorimotor training and thus improve treatment outcome. PURPOSE: To compare, in terms of symptoms, functional limitations and shoulder control, a group receiving a rehabilitation program centered on sensorimotor training combined with tDCS to a group receiving the same rehabilitation program combined with sham tDCS in individuals with RC tendinopathy. METHODS: Forty adults with RC tendinopathy will take part in the 4 evaluation sessions (0, 3, 6, 12 weeks) and a 6-week rehabilitation program. Outcome measures will be symptoms and functional limitations (Disability of the Arm, Shoulder and Hand and the Western Ontario Rotator Cuff index), as well as acromiohumeral distance ([AHD] ultrasonographic measurement at 0° and 60° of elevation arm). The rehabilitation program will include sensorimotor training, strengthening and education. tDCS will be apply during sensorimotor training on the motor cortex contralateral to the side of pain. A 2-way ANOVA will be used to analyse the effects of tDCS on the outcomes.

DETAILED DESCRIPTION:
BACKGROUND: tDCS is a safe and easy to use technique that has emerged as a promising tool to induce plasticity and to facilitate sensorimotor rehabilitation with potential application in various clinical populations. tDCS has been shown to induce changes that outlast the duration of the stimulation, by modulating neuronal membrane potential of the targeted brain region. Depending on the flow of current, tDCS can increase or decrease neuronal excitability; anodal tDCS induces membrane depolarization and enhanced excitability of cortical neurons, whereas cathodal tDCS induces membrane hyperpolarization and reduced excitability of cortical neurons. As such, tDCS has the potential to prime the plastic potential of a given brain region, making it more responsive to another intervention. For example, it has been shown that five days of anodal tDCS combined with training promotes motor skill acquisition still detectable three months later; an effect significantly superior to sham tDCS. These effects most likely are due to the augmentation of synaptic plasticity that requires the presence of brain-derived neurotrophic factor.

Coupled with sensorimotor training, tDCS can lead to subsequent sustained clinical gains.The beneficial effects of tDCS combined with sensorimotor training to normalize motor cortical activity and to enhance rehabilitation have been shown in populations with neurological injuries, such a stroke. In musculoskeletal populations, anodal tDCS over M1 has also been shown to lead to significant pain level reduction. Evidence suggests that tDCS over M1 may relieve pain through inhibition of thalamic sensory neurons and disinhibition of neurons located in the periaqueductal gray matter. In these latter studies, tDCS was specifically aimed at reducing pain and was not coupled with sensorimotor training. In fact, evidence on the effect of tDCS coupled with sensorimotor training in musculoskeletal populations is scarce, and the effect of such intervention has never been evaluated in individuals with RC tendinopathy. Considering that RC tendinopathy is associated with impaired motor control and that pain can decrease the excitability of the motor cortex and impair motor learning, the investigators believe that it is relevant to determine whether tDCS can enhance sensorimotor training, and improve outcome.

PURPOSE - The primary objective of this randomized control trial is to compare, in terms of symptoms and functional limitations, a group receiving a rehabilitation program centered on sensorimotor training combined with anodal tDCS to a group receiving the same rehabilitation program combined with sham tDCS in individuals with RC tendinopathy. A secondary objective is to explore the effects of these interventions on shoulder control and corticospinal excitability.

METHODS - Study Design: This triple-blind (patients, therapist & evaluator), parallel-group randomized control trial will include four evaluation sessions over 6 months (baseline, week 3, week 6, 3-month) and a 6-week rehabilitation program.

Interventions: Each participant will take part in the same 8-week rehabilitation program supervised by an independent physiotherapist. This program, previously shown effective, targets the deficits described in individuals with RC tendinopathy. It includes sensorimotor training, strengthening, and patient education. Each session lasts 40 minutes, with at least 75% for sensorimotor training. The rest of the session is used to teach and revise home exercises. tDCS will be applied during sensorimotor training (30 min),but only during the first five sessions, as these sessions will be during the first phase of motor learning, characterized by considerable improvement in performance.

Statistical Analyses - Descriptive statistics will be used for all outcome measures at each measurement time to summarise results. Baseline demographic data will be compared (independent t-test and Chi-squared tests) to establish the comparability of groups. All data will be tested to check the distributional assumptions for the inferential statistical analyses. An intention-to-treat analysis will be used in which all participants will be analysed in the group to which they were originally assigned. All dropouts and the reason for dropping out of the study will be reported. Any harm or unintended effects during the programs will be recorded. A 2-way ANOVA (2 tDCS [Real or Sham] x 4 Time [week 0, 3, 6, 12]) will be used to analyse the effects of tDCS on primary outcome and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* painful arc of movement
* positive Neer or Kennedy-Hawkins tests
* pain on resisted isometric lateral rotation or abduction, or positive Jobe test. The diagnosis accuracy of the combination of these tests has been studied (sensitivity & specificity ≥ 0.74)

Exclusion Criteria:

1. fracture at the symptomatic upper limb;
2. previous neck or shoulder surgery;
3. shoulder pain reproduced during active neck movement;
4. shoulder capsulitis;
5. clinical signs of a full thickness RC tear;
6. rheumatoid, inflammatory, or neurological diseases;
7. behavioural or cognitive problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Symptoms perceived at week 3,6 and 12. | At week 3, 6, and 12, the self-administered DASH questionnaires will be administered.
  Change from Baseline Symptoms perceived at week 3,6 and 12 with DASH (Disability of the Arm, Shoulder and Hand; self-administered questionnaire)
Change from Functional limitations perceived at week 3,6 and 12. | At week 3, 6, and 12, the self-administered WORC questionnaire will be administered.
  Change from Functional limitations at week 3,6 and 12 with WORC (Western Ontario Rotator Cuff Index; self-administered questionnaire)

SECONDARY OUTCOMES:
Change from US measurement of supraspinatus tendon at week 0 and 6. | US measurement will be performed at week 0 and 6.
  US measurement of supraspinatus tendon will be assessed. Supraspinatus tendon measures will be obtained with the transducer perpendicularly, one centimeter behind to the anterolateral aspect of the surface of the acromion. The thickness of the tendon borders will be defined inferiorly as the first hyperechoic region above the anechoic articular cartilage of the humeral head, and the hyperechoic superior border of the tendon before the anechoic subdeltoid bursa. Three measures will be taken, and the mean tendon thickness measured will be expressed as a percentage of the mean AHD at rest using the following formula: occupation ratio = [(tendon thickness/AHD) x 100].
Change from Corticospinal excitability of the infraspinatus (IS) muscle at day 1 before the first treatment and day 1 after the first treatment. | Through first tDCS treatment of each participant.
  Corticospinal excitability of the infraspinatus (IS) muscle will be acquired using a stimulator. Stimuli will be applied over grid sites spaced 1 cm apart and positioned over the upper limb area of primary motor cortex (M1). Prior to the experiment, subjects will be asked to perform two IS maximal voluntary contractions (MVC). Maximal value over the two trials will be used to compute electromyographic targets during experimental task. Corticospinal excitability will be evaluated during slight voluntary contraction.The optimal location for stimulation of IS will be determined (hotspot), as well as the active motor threshold (aMT) at this site. aMT will be determined as the minimal intensity of stimulation required to elicit motor evoked potential (MEP) larger than 150 μ Volts in at least 6 out of 12 trials at the hotspot for IS at 5% of MVC. Ten stimulations will be performed at the hotspot at 120% of the threshold for IS.
Change from US measurement of AHD at week 0 and 6. | US measurement of AHD will be performed at week 0 and 6.
  US measurement of AHD will be performed using an ultrasound scanner with a 7.5-12 Mhz linear array probe. The US measurement of AHD is defined as the tangential distance between the hyperechoic bony landmarks of the humeral head and the inferior edge of the acromion visible on the longitudinal sonogram. Measurement obtained represents the AHD at the anterior outlet of the subacromial space. Measurements will be taken in a sitting position with the arm at rest, and at 45° and 60° of active abduction. For each arm position, two measures will be taken, and the mean AHD will be calculated. These measures are highly reliable (ICC > 0.90).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, Pht,PhD, Study Director — Center of Interdisciplinary Research in Rehabilitation and Social Integration, Quebec City, Laval University, Quebec City, Canada
Locations (1):
- Center of Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The data of the acromio-humeral distance could be shared with a group of students who will work on a systematic review (group with pain vs. control group).

REFERENCES:
- [Background] Roy JS, Moffet H, McFadyen BJ. Upper limb motor strategies in persons with and without shoulder impingement syndrome across different speeds of movement. Clin Biomech (Bristol). 2008 Dec;23(10):1227-36. doi: 10.1016/j.clinbiomech.2008.07.009. Epub 2008 Aug 30. PMID 18757123
- [Background] Ngomo S, Mercier C, Bouyer LJ, Savoie A, Roy JS. Alterations in central motor representation increase over time in individuals with rotator cuff tendinopathy. Clin Neurophysiol. 2015 Feb;126(2):365-71. doi: 10.1016/j.clinph.2014.05.035. Epub 2014 Jun 21. PMID 25043198
- [Background] Tsao H, Galea MP, Hodges PW. Driving plasticity in the motor cortex in recurrent low back pain. Eur J Pain. 2010 Sep;14(8):832-9. doi: 10.1016/j.ejpain.2010.01.001. Epub 2010 Feb 23. PMID 20181504
- [Background] Desmeules F, Minville L, Riederer B, Cote CH, Fremont P. Acromio-humeral distance variation measured by ultrasonography and its association with the outcome of rehabilitation for shoulder impingement syndrome. Clin J Sport Med. 2004 Jul;14(4):197-205. doi: 10.1097/00042752-200407000-00002. PMID 15273525
- [Background] Roy JS, Moffet H, Hebert LJ, Lirette R. Effect of motor control and strengthening exercises on shoulder function in persons with impingement syndrome: a single-subject study design. Man Ther. 2009 Apr;14(2):180-8. doi: 10.1016/j.math.2008.01.010. Epub 2008 Mar 20. PMID 18358760
- [Background] Vaseghi B, Zoghi M, Jaberzadeh S. Does anodal transcranial direct current stimulation modulate sensory perception and pain? A meta-analysis study. Clin Neurophysiol. 2014 Sep;125(9):1847-58. doi: 10.1016/j.clinph.2014.01.020. Epub 2014 Feb 4. PMID 24555922
- [Background] Feng WW, Bowden MG, Kautz S. Review of transcranial direct current stimulation in poststroke recovery. Top Stroke Rehabil. 2013 Jan-Feb;20(1):68-77. doi: 10.1310/tsr2001-68. PMID 23340073
- [Background] Siebner HR, Lang N, Rizzo V, Nitsche MA, Paulus W, Lemon RN, Rothwell JC. Preconditioning of low-frequency repetitive transcranial magnetic stimulation with transcranial direct current stimulation: evidence for homeostatic plasticity in the human motor cortex. J Neurosci. 2004 Mar 31;24(13):3379-85. doi: 10.1523/JNEUROSCI.5316-03.2004. PMID 15056717